CLINICAL TRIAL: NCT03110432
Title: Prospective German Very High Cardiovascular Risk Patients Dyslipidemia Treatment Indication Registry
Acronym: PERI-DYS
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: PERI-DYS
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Dyslipoproteinemias; Hypercholesterolemia, Familial; Familial Hypercholesterolemia - Homozygous; Familial Combined Hyperlipidemia
Keywords: Cardiovascular; LDL Cholesterol; Drug utlisation; high risk; secondary prevention; PCSK9 inhibition
MeSH Terms: conditions — Dyslipidemias; Hyperlipoproteinemia Type II; Homozygous Familial Hypercholesterolemia; Hyperlipidemia, Familial Combined | interventions — erucylphosphocholine; evolocumab; alirocumab; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Niacin; Fibric Acids; Colesevelam Hydrochloride; Fatty Acids, Omega-3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard lipid lowering therapy: Statins, ezetimibe, nicotinic acid, fibrates, cholestagel, omega-3 fatty acids (and any combinations of these agents)
  Interventions: Drug: Standard lipid lowering therapy
- PCSK9 Inhibitor [EPC]: Evolocumab or alirocumab.
  Interventions: Drug: PCSK9 Inhibitor [EPC]

INTERVENTIONS:
Drug: PCSK9 Inhibitor [EPC] — drug use according to the respective product labelling
  Other Names: Repatha, Praluent
  Groups: PCSK9 Inhibitor [EPC]
Drug: Standard lipid lowering therapy — drug use according to the respective product labelling
  Other Names: Statins, ezetimibe, nicotinic acid, fibrates, cholestagel, omega-3 fatty acids
  Groups: Standard lipid lowering therapy

SUMMARY:
This is a prospective German registry for patients with dyslipidemia with very high cardiovascular risk who principally meet the Gemeinsamer Bundesausschuss (G-BA) stipulations for Proprotein convertase subtilisin/kexin like type 9 inhibitor (PCSK9i) use, and are treated by office-based cardiologists or in lipid ambulances.

DETAILED DESCRIPTION:
The study is purely observational, and will document data from the patient charts only. Treatment of patients will not be changed by this study, and all clinical decisions (including on frequency of visits) will be upon the discretion of the physician. No blood samples must be taken solely for the purpose of the study.

The registry will include two types of centers: 1) office-based cardiologists and 2) specialized lipid ambulances (outpatient departments).

Data on patient disease and treatment history will be collected a first documentation (retrospectively).

The documentation time is 3 years per patient. After the baseline visit, patients are followed-up every 6 ± 2months (last visit at month 36). This interval is considered narrow enough not to miss important events (safety reporting, cardiovascular events, hospitalizations).

Patients with stable (maintenance) lipid-lowering therapy (including those with existing PCSK9i therapy) or those with any therapy changes (including newly initiated PCSK9i treatment) will be documented in this study. Compared to the former group with stable drug treatment, the latter group will likely have major LDL-C changes during the first few weeks, which will be accounted for by (retrospective) monthly documentation in the first 3 months (data will be documented at the 6-month visit.

The documentation periods will be substantially longer than in the controlled studies of the PCSK9i (endpoints were as early as 3 months), and thus will provide much-needed information about the long-term effects on LDL-C and other lipid parameters, safety, and drug retention rates. Longer follow-up periods would likely be compromised by high rates of (administrative) discontinuation rates.

ELIGIBILITY:
Inclusion Criteria:

* • with familial, homozygous hypercholesterolemia, in whom pharmaceutical and diet options for lipid lowering have proved insufficient, or

  * with confirmed familial, heterozygous hypercholesterolemia under consideration of the total familial risk, or
  * with heterozygous familial or non- familial hypercholesterolemia or mixed dyslipidemia with

    * therapy refractory course
    * maximal dietary and pharmaceutical lipid lowering therapy - in any case documented over a 12-month period
    * unsatisfactorily lowered LDL-C value (and thus with an indication for LDL apheresis)
    * confirmed vascular disease
    * other risk factors for cardiovascular events

Exclusion Criteria:

* Concurrent participation of the patient in a clinical randomised study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyslipidemia and very high cardiovascular risk ("highest risk patients" according to G-BA stipulation for PCSK9i use)
Sampling Method: Non-Probability Sample
Enrollment: 1695 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol goal achievement | 3 years
  < 70 mg/dl

SECONDARY OUTCOMES:
LDL cholesterol reduction | up top 3 years
  Compared to baseline
Number of treatment changes | up to 3 years
  During the follow-up period

OTHER OUTCOMES:
Change in quality of life | up to 3 years
  by EuroQol 5 dimensions

CONTACTS AND LOCATIONS:
Overall Officials: David Pittrow, MD, PhD, Principal Investigator — GWT-TUD GmbH, Germany; Andreas Birkenfeld, MD, PhD, Study Chair — Innere Medizin IV - Diabetologie, Endokrinologie und Nephrologie am Universitaetsklinikum Tuebingen, Germany; Bernd Hohenstein, MD, PhD, Study Chair — Nephrologisches Zentrum Villingen-Schwenningen, Germany; Ulrich Laufs, MD, PhD, Study Chair — Klinik für Innere Medizin III, Universität des Saarlandes, Germany; Volker JJ Schettler, MD, PhD, Study Chair — Nephrologisches Zentrum Göttingen GbR, Germany; Elisabeth Steinhagen-Thiessen, MD, PhD, Study Chair — Lipid Clinic, Charité Universitaetsmedizin, Berlin, Germany; Klaus G Parhofer, MD, PhD, Study Chair — Ludwig Maximilian University, Medizinische Klinik und Poliklinik IV, Muenchen, Germany
Locations (3):
- Germany (3):
  - Klinik und Poliklinik für Kardiologie, Universitätsklinikum, Leipzig
  - Innere Medizin IV - Diabetologie, Endokrinologie und Nephrologie am Universitaetsklinikum, Tübingen
  - Nephrologisches Zentrum, Villingen-Schwenningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parhofer KG, Pittrow D, Birkenfeld AL, Fraass U, Hohenstein B, Siegert C, Klotsche J, Steinhagen-Thiessen E, Dexl S, Schettler VJJ, Laufs U. Determinants of lipid lowering therapy intensification in very high risk patients with dyslipidaemia eligible for PCSK9 monoclonal antibodies: 1-year outcomes of the PERI-DYS study. Acta Cardiol. 2025 Jul;80(5):475-486. doi: 10.1080/00015385.2025.2490381. Epub 2025 Apr 24. PMID 40270128
- [Background] Laufs U, Birkenfeld AL, Fraass U, Hohenstein B, Siegert C, Klotsche J, Steinhagen-Thiessen E, Pittrow D, Dexl S, Salmen S, Schettler VJJ, Parhofer KG; Collaborators in the PERI-DYS Study. Novel Insights into the Management of Patients with Very High Cardiovascular Risk Eligible for PCSK9 Inhibitor Treatment: Baseline Findings from the PERI-DYS Study. Cardiovasc Drugs Ther. 2024 Feb;38(1):119-129. doi: 10.1007/s10557-022-07386-0. Epub 2022 Sep 30. PMID 36178485
- [Derived] Parhofer KG, Pittrow D, Birkenfeld AL, Fraass U, Hohenstein B, Siegert C, Klotsche J, Steinhagen-Thiessen E, Dexl S, Schettler VJJ, Laufs U. Treatment persistence, lipid lowering, and 3-year clinical outcomes in patients at very high cardiovascular risk on PCSK9 monoclonal antibodies. Clin Res Cardiol. 2026 Feb;115(2):288-303. doi: 10.1007/s00392-025-02719-z. Epub 2025 Aug 4. PMID 40760109